CLINICAL TRIAL: NCT00166673
Title: A Pilot Study to Evaluate the Navigator Continuous Glucose Sensor in the Management of Type 1 Diabetes in Children
Brief Title: Pilot Study of the Navigator Continuous Glucose Monitor
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: DirecNet 006; HD041890; HD041919; HD041908; HD041906; HD041918; HD041915
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: Diabetes Mellitus, Insulin-Dependent; Type 1 Diabetes; Continuous Glucose Monitoring Devices; Electronic Data Collection
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Device: FreeStyle Navigator Continuous Glucose Monitoring System

SUMMARY:
This study is being done to find out how accurate the Navigator continuous glucose monitor is in children. It is also being done to see if use of the Navigator can improve blood sugar control and help prevent low blood sugar events. This study has three basic parts: Use of the Navigator at home for one week without being able to see the blood sugar readings; a Baseline visit or a 24-hour admission to a research unit of the hospital to find out how well the Navigator measures the blood sugar; and then 3 months use of the Navigator at home as an aid to diabetes care.

DETAILED DESCRIPTION:
Approximately 60 children will be recruited from five centers in the United States to participate in this study. The information gained from this study will be used to plan a larger study in which half of the patients will use the Navigator and half will not. Children who participate in this study will not be eligible to take part in the larger study.

The Navigator provides a glucose reading every 60 seconds (or 1440 readings a day). Each sensor is designed to provide readings for up to 120 hours. It has alarms for hypoglycemia and hyperglycemia and for projected high and low glucose values. The alarm set points can be adjusted by the user. The Navigator also has a trend arrow indicating the glucose rate of change (>-2 mg/dL/min, -2 to -1 mg/dL/min, -1 to 1 mg/dL/min, 1 to 2 mg/dl/min, and >2 mg/dl/min). Subjects can enter events, such as when they took insulin, ate, or exercised. The sensor requires calibration values to be entered 3 times during the first day of wear at 1-hour, 3-hours, and 24-hours and does not require additional calibration values. The values are entered directly into the Navigator which has a TheraSense Freestyle home glucose meter built into the unit. The Navigator has not yet been approved by the FDA. The Navigator currently under review by the FDA will limit sensor wear to 3 days.

Beginning the Study

When a child enters the study, the following will be done:

1. Questionnaires will be completed.

   * Parents and children (if at least 9 years old) will be asked to fill out questionnaires on a computer in the clinic. The questions will be about the child's diabetes, how the diabetes is being treated, and how the diabetes affects the parent and child.
   * Children who are using insulin pump therapy and are at least 9 years old and parents will be interviewed about the child's diabetes management habits at home. The interview will be conducted by phone by trained interviewers who are at Nemours Children's Clinic in Jacksonville, Florida, one of the study sites.
2. Blood will be drawn to measure glycosylated hemoglobin (HbA1c).
3. Parents and children will be instructed on using the Navigator. The first sensor will be inserted by the parent or child with guidance from the study nurse. During the first week, the parent and child will not be able to see the results from the Navigator.
4. Children will be asked to do the following before returning for the Baseline Visit or the hospital stay about 1 week later:

   * Check the blood sugar using the Freestyle meter built into the Navigator at least 4 times a day
   * Wear the Navigator sensor everyday and change the sensor at the end of day 5
   * On the day a new sensor is started, do 3 fingerstick blood sugar readings using the built-in Freestyle meter to calibrate the Navigator
   * Enter a meal marker event into the Navigator each time your child has a meal or snack
   * Insert a new sensor 1, 2, 3, or 4 days before your child will stay in the hospital
   * Bring any used sensors, including the packaging and inserting device to the Baseline Visit or hospital stay

Baseline Visit Children who are using Lantus with MDI therapy will return for a Baseline Visit approximately one week (7-12 days) after the enrollment visit.

Hospital Stay Those children who are using insulin pump therapy will return for a hospital stay approximately one week (7-12 days) after the enrollment visit and will use the Navigator for about 24 hours. The last sensor that was placed at home will continue to be worn during the hospital stay. A new sensor will also be placed so that your child has 2 sensors inserted during the hospital stay to see how closely the 2 sensors agree.

A CGMS sensor will be inserted and calibrated one hour later.

A small tube called a catheter will be placed in a vein in the child's arm and will stay in the vein while the child is in the hospital. From this tube, a very small blood sample will be drawn every 30 minutes during the hospital stay. After breakfast, blood samples will be taken about every 10 minutes for about an hour. For children who are at least 7 years old, blood samples will be taken about every 20 minutes during a period of exercise in the afternoon.

Procedures at Home after the Baseline Visit or Hospital Stay

1. Use the Navigator.

   * The Navigator should be worn all of the time for 3 months.
   * The sensor must be replaced every 5 days.
   * With each sensor wear 4 blood sugar readings must be done using the built-in Freestyle meter to calibrate the Navigator.
   * Enter a meal marker event into the Navigator each time a meal or snack is eaten.
   * Children may be asked to insert a new sensor 5 days before some of the study visits to allow the study personnel to look at the skin after the sensor has been worn for 5 days.
2. Download the Navigator - Once a week, children will need to download the glucose results from the Navigator, which will then be emailed to the study coordinating center.
3. Use Algorithms for Diabetes Management Decisions - The study doctor or nurse will give the parents and children instructions (Algorithms) for how to make changes to diabetes management from the results of the Navigator. The instructions will be used by the parents and children to make decisions as they receive the results from the device.
4. Phone Interviews - After 3 days and 2, 4, 8, and 10 weeks after the children leave the hospital, one of the staff will call to see how they is doing with the Navigator and the instructions for diabetes management decisions. We will ask what the child ate in the last meal before the call. We also will ask if the child has been sick or under any stress. For females who have started menstruating, we will ask about her menstrual cycle.

Study Visits

Children will return to the diabetes clinics for visits 1, 3, 7, and 13 weeks after the hospital stay. At these visits, the following will be done:

1. Any used sensors, including the packaging and inserting device will be collected.
2. The skin will be looked at where the Navigator has been worn.
3. The Navigator and the child's insulin pump will be downloaded and reviewed with the parent and child.
4. The diabetes management instructions will be reviewed with the parent and child to determine if the instructions have been helpful or if they need to be changed.

At the 3, 7, and 13- week visits, parents and children (if at least 9 years old) will be asked to complete a questionnaire about how much you liked or disliked the instructions that were given for using the results of the Navigator.

At the 7-week visit, the following will also be done in addition to the child's regular clinic visit:

1. Blood will be drawn to measure the HbA1c.

At the 13-week visit, the following will also be done in addition to the child's regular clinic visit:

1. Blood will be drawn to measure the HbA1c.
2. Questionnaires will be completed

   * Parents and children (if at least 9 years old) will be asked to complete the same questionnaires and the phone interview that were done during the first visit.
   * Parents and children will be asked to complete one more questionnaire about how much they like using the Navigator.
3. If the children are willing to continue using the Navigator, they will be given additional sensors to use as often as they would like and they will return for another regular clinic visit in about 3 months (26-week visit). At that visit, the skin will be looked at where the Navigator was used, the HbA1c will be measured, and the parents and children will be asked to complete the same questionnaires that were completed at the 13-week visit about how much they liked using the Navigator and the instructions that were given for using the results of the Navigator.

Those who decide to continue using the Navigator will be seen again at 26-weeks.

* At the 26-week visit, subjects will be given the choice to continue in the study until the device is approved by the FDA or until Abbott Diabetes Care can no longer provide supplies for the study. Subjects who agree to continue in the study will sign an addendum to the informed consent.
* Subjects who continue in the study will return to the clinic every 3 months for a follow-up visit. The same procedures completed during the 26-week visit will be completed at each subsequent visit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
* Age 3.0 years to less than 18.0 years
* Subject has used a downloadable insulin pump or Lantus with MDI of a short-acting insulin (e.g. Humalog or Novolog) for at least 6 months
* Parent/guardian and subject understand the study protocol and agree to comply with it
* Subjects >9.0 years old and primary care giver (i.e., parent or guardian) comprehend written English
* Subject has a home computer with email access
* For females, subject not intending to become pregnant during the next 3 months
* No expectation that subject will be moving out of the area of the clinical center during the next 3 months
* Informed Consent Form signed by the parent/guardian and Child Assent Form signed by the subject

Exclusion Criteria:

* The presence of a significant medical disorder that in the judgment of the investigator will affect the wearing of the sensors or the completion of any aspect of the protocol.
* The presence of any of the following diseases:

  * Asthma if treated with systemic or inhaled corticosteroids in the last 6 months
  * Cystic fibrosis
  * Other major illness that in the judgment of the investigator might interfere with the completion of the protocol (Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment)
* Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian).
* Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2005-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of using the Navigator sensor on a daily basis (Average number of sensors used per week, Average number of hours of use per sensor, Number of sensors per week that fail to calibrate)
Navigator Accuracy

SECONDARY OUTCOMES:
Psychosocial Questionnaires
Exploratory assessment of impact of Navigator on HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: William V Tamborlane, M.D., Study Chair — Yale University
Locations (6):
- United States (6):
  - Division of Pediatric Endocrinology and Diabetes, Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Aurora, Colorado
  - Department of Pediatrics, Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jaeb Center for Health Research, Tampa, Florida
  - Department of Pediatrics, University of Iowa Carver College of Medicine, Iowa City, Iowa

REFERENCES:
- [Result] Buckingham B, Ruedy K, Kollman C, Beck R, Tamborlane W, Mauras N, Weinzimer S, Chase P, Tsalikian E; and the Diabetes Research in Children Network (DirecNet) Study Group. Family Assessment of the Utility of the DirecNet Applied Treatment Algorithm (DATA) for Insulin Adjustments in Real-Time and Retrospective Analyses of Continuous Glucose Monitoring (CGM) Diabetes 2006; 55(Suppl.1): A453
- [Result] Fiallo-Scharer R, Tamborlane W, Buckingham B, Wysocki T, Weinzimer S, Tsalikian E, Beck R, Ruedy K, Kollman C; and the Diabetes Research in Children Network (DirecNet) Study Group. Diabetes Research in Children Network (DirecNet) Pilot Study to Evaluate the FreeStyle Navigator® Continuous Glucose Monitoring System in the Management of T1D in Children. Diabetes 2006; 55(Suppl.1): A452.
- [Result] Wilson DM, Beck RW, Tamborlane WV, Dontchev MJ, Kollman C, Chase P, Fox LA, Ruedy KJ, Tsalikian E, Weinzimer SA; DirecNet Study Group. The accuracy of the FreeStyle Navigator continuous glucose monitoring system in children with type 1 diabetes. Diabetes Care. 2007 Jan;30(1):59-64. doi: 10.2337/dc06-1407. PMID 17192334
- [Result] Diabetes Research in Children Network (DirecNet) Study Group. Relative accuracy of the BD Logic and FreeStyle blood glucose meters. Diabetes Technol Ther. 2007 Apr;9(2):165-8. doi: 10.1089/dia.2006.0005. PMID 17425442
- [Result] Diabetes Research in Children Network (DirecNet) Study Group; Buckingham B, Beck RW, Tamborlane WV, Xing D, Kollman C, Fiallo-Scharer R, Mauras N, Ruedy KJ, Tansey M, Weinzimer SA, Wysocki T. Continuous glucose monitoring in children with type 1 diabetes. J Pediatr. 2007 Oct;151(4):388-93, 393.e1-2. doi: 10.1016/j.jpeds.2007.03.047. Epub 2007 Aug 24. PMID 17889075
- [Result] Messer L, Ruedy K, Coffey J, Englert K, Caswell K, Steffen A; and the Diabetes Research in Children Network (DirecNet) Study Group. Pediatric Educators' Role in Successful Continuous Glucose Monitoring. Diabetes 2007; 56(Suppl.1): A617.
- [Result] Diabetes Research In Children Network (DirecNet) Study Group; Buckingham B, Xing D, Weinzimer S, Fiallo-Scharer R, Kollman C, Mauras N, Tsalikian E, Tamborlane W, Wysocki T, Ruedy K, Beck R. Use of the DirecNet Applied Treatment Algorithm (DATA) for diabetes management with a real-time continuous glucose monitor (the FreeStyle Navigator). Pediatr Diabetes. 2008 Apr;9(2):142-7. doi: 10.1111/j.1399-5448.2007.00301.x. Epub 2008 Jan 24. PMID 18221427